CLINICAL TRIAL: NCT04141215
Title: Allogeneic Bone Paste Versus Allogeneic Bone Powder in Pre-implant Guided Bone Regeneration in Oral Surgery: a Randomized Non-inferiority Clinical Trial
Brief Title: Allogeneic Bone Paste Versus Allogeneic Bone Powder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biobank (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-A00488-49
Record Dates: First submitted 2019-10-23; First posted 2019-10-28 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-01

CONDITIONS: Bone Resorption; Dental Diseases
MeSH Terms: conditions — Bone Resorption; Stomatognathic Diseases

STUDY DESIGN:
Intervention Model Description: Randomized non-inferiority, two-arm, parallel, single-blind and monocentric clinical trial:
  1. BIOBank bone paste (PPT322), derived from human living donor femoral heads
  2. BIOBank cortico-cancellous bone powder (PPT6), derived from human living donor femoral heads, used in current practice as reference treatment
Who Masked: Participant, Outcomes Assessor
Masking Description: Statistician will also perform trial analyses with treatment masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIOBank bone paste (PPT322) (Experimental): Allogeneic bone paste derived from human living donor femoral heads
  Interventions: Biological: BIOBank bone paste
- BIOBank cortico-cancellous bone powder (PPT6) (Active Comparator): Allogeneic bone powder derived from human living donor femoral heads (used in current practice)
  Interventions: Biological: BIOBank cortico-cancellous bone powder

INTERVENTIONS:
Biological: BIOBank bone paste — BIOBank bone paste (PPT322)
  Arms: BIOBank bone paste (PPT322)
Biological: BIOBank cortico-cancellous bone powder — BIOBank cortico-cancellous bone powder (PPT6)
  Arms: BIOBank cortico-cancellous bone powder (PPT6)

SUMMARY:
Autogenous bone graft has been considered the gold standard in Guided Bone Regeneration (GBR) technique used for bone augmentation. However, there are disadvantages associated with autograft use such as limited amount of available bone and increased morbidity for the patient at the sampling site. Several biomaterials have been used as a replacement of the autogenous bone. Viral-inactivated bone allograft powder is an alternative that has proven efficacy and tolerance. This study aims to assess the non-inferiority of viral-inactivated allogeneic bone paste compared to a viral-inactivated cortico-cancellous allogenic bone powder in achieving the ideal bone volume.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged ≥ 18 years old
2. Patient able to read, understand and give written consent to participate in the study
3. Patient affiliated with a social security system or beneficiary of such a system
4. Partially edentulous patient with 1 to 2 intercalary missing teeth or a terminal gap with distal vertical and lateral support bone volume
5. Presence of a bone deficit requiring horizontal and / or vertical bone augmentation (stage 4 or 5 of the Benic and Hammerle classification) treated by GBR for delayed placement of up to 4 dental implants
6. Possibility of acquisition by CBCT for the required protocol visits

Exclusion Criteria:

1. General contraindication to bone graft and implant surgery
2. Pregnant woman or planned pregnancy during the study period or breast-feeding woman;
3. Patient who has had a bone augmentation by GBR during the previous 12 months, in the area targeted for filling with the allogeneic material
4. Patient who received less than 3 months ago a CBCT acquisition at the operative site
5. Patient simultaneously requiring more than one GBR augmentation in the same quadrant
6. Patient with signs of local infection at the targeted graft site
7. Systemic, metabolic or autoimmune disease that may adversely affect healing of soft and bone tissue (eg, unbalanced type 1 or type 2 diabetes)
8. Use of treatments (chemotherapy or radiotherapy) or drugs (bisphosphonates, chronic steroids) known to potentially interfere with tissue healing
9. Patient presenting a dental plaque objectified by an oral examination (Loe SILNESS ≥ 2 on more than 50% of the dental surfaces)
10. Patient smoker of more than 10 cigarettes a day
11. Any other condition that, in the investigator's opinion, would be detrimental to the safety of the patient or fail to meet the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Bone volume obtained | 4 to 6 months post-bone grafting
  The primary endpoint is binary in nature (yes / no) and assessed radiographically by the CBCT: To assess, 4 to 6 months post-transplant, if the bone volume obtained at the time of implant placement corresponds to the desired bone volume before the transplant.
  Measured by an independent Evaluator, blind to the treatment received.

SECONDARY OUTCOMES:
Duration of surgery | immediate post-operative
  measured in minutes
Ease of manipulation | immediate post-bone grafting
  assessed by the operating surgeon using a Visual Analogue Scale from 0 (Not easy at all) to 10 (Very easy)
Absolute gain in bone volume | 4 months post-bone grafting
  measured in mm by a radiographic distance
Primary osteointegration (implants stability) | 4 months post-bone grafting
  measured by Implant Stability Quotient (ISQ) using Resonance frequency analysis (RFA)
Peri-implant marginal bone height | 4 months post-bone grafting
  measured in mm
Survivorship of the implant | 3-4 months post-implant
  binary variable yes / no
Need for a new bone augmentation simultaneously with implant placement | 4 to 6 months post-bone grafting (implant placement)
  Binary yes/no
Insufficient primary stability of the implant | 4 to 6 months post-bone grafting (implant placement) and 3-4 months post-implant
  Implant Stability Quotient (ISQ) less than 35N
Occurrence of complications related to the transplant | 7-10 months post-bone grafting
  binary yes / no
Nature of possible complications or a thematic grouping in the inter-group comparison | 7-10 months post-bone grafting
  All complications appeared from the bone grafting until the end of the study will be described overall and by arm and grouped by thematic if relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Courtois, Dr, Principal Investigator — Clinique Rive Gauche (TOULOUSE)
Locations (1):
- Clinique Rive Gauche, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Courtois B, L'Homme A, Labadie MP. Allogeneic bone paste versus bone powder for oral guided bone regeneration: A randomized, noninferiority trial. J Periodontol. 2025 Oct 29. doi: 10.1002/jper.11385. Online ahead of print. PMID 41159915